CLINICAL TRIAL: NCT03621306
Title: Precision and Reliability of Dual X-ray Absorptiometry (DXA) Testing
Brief Title: DXA Study of Precision and Reliability
Status: Recruiting | Type: Observational
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Mary Jane DeSouza, Professor of Kinesiology, Penn State University
Other Study IDs: DXAPrecision
Record Dates: First submitted 2018-08-03; First posted 2018-08-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Bone and Bones; Body Composition
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Men and women aged 18+: Men and women over the age of 18
  Interventions: Device: DXA and pQCT precision testing

INTERVENTIONS:
Device: DXA and pQCT precision testing — The participants are only being observed; there is no intervention other than DXA and pQCT testing for the purposes of looking at instrument/technician precision..

SUMMARY:
The purpose of the study is to assess precision of the GE Lunar iDXA, Hologic Horizon W DXA scanner, and the Stratec peripheral quantitative computed tomography (pQCT) scanner.

Aim 1: To assess standard deviation (SD) and coefficient of variation (CV) of testing bone mineral, bone geometry, and soft tissues in inanimate objects and adults. Tests on adults will be structured to assess:

1. Within- and between-day variability of testing
2. Within- and between-technician variability of testing
3. Variability due to positioning and post-scan processing
4. Variability due to different DXA scanning equipment

Aim 2: To assess the least significant change (LSC) for testing bone mineral and soft tissues in adults.

Aim 3: To assess strengths and limitations of DXA and pQCT testing, including sensitivity to movement, rate of re-rescanning, etc. which are crucial components for demonstrating feasibility in grant applications.

Aim 4: To construct a database of DXA and pQCT test results and quality control procedures, showing our laboratory's quality control level.

DETAILED DESCRIPTION:
Osteoporosis and obesity are highly prevalent and disabling chronic diseases. Osteoporosis is a disease of low bone mass, which predisposes people to bone fragility and increased risk of bone fractures. Obesity is a disease characterized by excess body fat levels, which predisposes people to diabetes, heart disease, stroke, hypertension, cancer, sleep apnea, osteoarthritis, and gallbladder disease.

An essential component to research on the prevention and treatment of osteoporosis and obesity is a valid method for monitoring body fat levels and bone mineral density. Dual energy X-ray absorptiometry (DXA) is a method for analyzing bone mineral density and body composition, particularly bone mineral content, fat mass and lean mass in children and adults. DXA scanners use an X-ray tube to produce radiation, which is then filtered into low- and high-energy beams. These beams of radiation are emitted from beneath a table that the supine human body is lying on. The arm, which passes above the person, detects the attenuation of the radiation for each pixel the body occupies. Based on known attenuation levels of different human tissues, the imaging software provides information on the composition of each pixel of the body. These pixels are then summed to provide information on: total body bone mineral content, total bone mineral density, fat mass, and lean mass. The DXA can also assess regional body composition (e.g. trunk fat), which is of importance in evaluating health effects of body fatness patterns. Using standard protocols, bone mineral content and density can be assessed in areas of the body indicating high risk of fractures (e.g. hip and lumbar spine) or areas that are likely to be responsive to dietary or physical activity manipulations (e.g. lumbar spine and radius).

Peripheral quantitative computed tomography (pQCT) is a 3-dimensional imaging technique that goes beyond the 2-dimensional imaging of DXA to assess both true volumetric bone density and bone geometry, the two key components of bone strength. Additionally, it can divide bone into its component parts, i.e. separately assessing bone density and bone geometry of cortical and trabecular bone. As such, the measurements obtained from pQCT provides a more complete picture of what may be occurring within bone tissue that contributes to either bone gain or bone loss, depending on the population and question of interest. pQCT assesses parameters of bone strength at the radius (forearm) and tibia (lower leg).

A vital component of any clinical and research program is precision testing, which assesses the reproducibility of DXA and pQCT measurements within an individual technician and/or between multiple technicians. This study was designed to address our facility's needs and ethical requirement to complete precision testing. This precision testing is a necessary component of verifying the feasibility and validity of the method, as well as cross-calibrating DXA scanners in our multi-site studies. We are completing this testing with the two DXA scanners, the GE Lunar iDXA and the Hologic Horizon W DXA, as well as with the Stratec XCT 3000 pQCT.

A vital component of any clinical and research program is precision testing, which assesses the reproducibility of DXA measurements within an individual technician and/or between multiple technicians. As alluded to above, the validity of bone and soft tissue measurements by DXA and pQCT is related to the skill of the technician in: 1) properly positioning the person before scanning and 2) properly analyzing the scan images afterward. Both of these components are subjective, requiring experience and feedback to improve technique.

From an ethical standpoint, a level of technician competency is important in ensuring that both research volunteers and the technician are not exposed to radiation without the benefit of acceptable scan results. From a clinical and research standpoint, understanding the inherent variability in testing is an important component in planning and executing research studies having bone or body fat outcomes. As described the Conference of Radiation Control Program Directors, Inc. (CRCPD), and as established by the International Society of Bone Densitometry (ISCD), measurement of precision is a key component for assessing:

1. The smallest change (least significant change, LSC) in bone density that is biologically significant
2. The time interval between measurements necessary to detect changes.

Precision testing requires that multiple scans be completed on individuals representative of the primary target population of interest, sometimes within a fairly short period of time. This exposure of additional radiation to a select group of individuals has created controversy about whether precision testing is necessary and ethical. The CRCPD and ISCD has fully supported precision testing, and recommended that it be a routine practice in all DXA sites. The CRCPD states that, "Some states without understanding the need for precision testing have prohibited the measurement despite low radiation doses and limited numbers of repeat densitometry determinations. Their major concern, of course, is the apparent unnecessary radiation to a few, select patients. To address the benefit versus risk issue, those exposed to the additional, small amount of radiation (equal to approximately an additional 6-12 hours of background radiation) are providing a benefit to themselves and all others by validating the results of bone mineral density (BMD) exams for that facility. Without precision testing, the BMD study is of no value resulting in thousands of patients being exposed to unnecessary radiation."

ELIGIBILITY:
Inclusion Criteria:

Healthy adults of two age groups, 1) aged 18-40 or 2) aged >40yr.

Exclusion Criteria:

1. for females, being pregnant
2. Having had X-ray procedures using contrast material in the previous 3 days
3. Having medical devices that interfere with scan accuracy
4. Wearing external metal objects that cannot be removed
5. Having internal metal objects
6. Body mass of > 450 lbs.
7. Having ostomies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will include men and women of all ages. Women must not be pregnant.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-06-16 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Precision of iDXA BMD | One month
  Standard Deviation and coefficient of variation for BMD measurements obtained on the GE Lunar iDXA
Precision of Hologic Horizon W DXA BMD | One month
  Standard Deviation and coefficient of variation for BMD measurements obtained on the Hologic Horizon W
Precision of iDXA Body Composition | One month
  Standard Deviation and coefficient of variation for body composition measurements obtained on the GE Lunar iDXA
Precision of Hologic Horizon W DXA Body Composition | One month
  Standard Deviation and coefficient of variation for body composition measurements obtained on the Hologic Horizon W
Precision of the Stratec XCT 3000 pQCT | One month
  Standard deviation and coefficient of variation for bone density, geometry, and estimated bone strength for the Stratec XCT 3000 pQCT

SECONDARY OUTCOMES:
LSC for the iDXA BMD | One month
  Least significant change for BMD using the GE Lunar iDXA
LSC for the Hologic Horizon W BMD | One month
  Least significant change for BMD using the Hologic Horizon W DXA
LSC for the iDXA body composition | One month
  Least significant change for body composition using the GE Lunar iDXA
LSC for the Hologic Horizon W body composition | One month
  Least significant change for body composition using the Hologic Horizon W DXA
LSC for the Stratec XCT 3000 | One month
  Least significant change for bone density, geometry, and estimated bone strength for the Stratec XCT 3000

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane De Souza, PhD, Principal Investigator — Penn State
Locations (1):
- Women's Health and Exercise Laboratories, The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No